CLINICAL TRIAL: NCT06630325
Title: Serial Measurements of Molecular and Architectural Responses to Therapy (SMMART): Adaptive Clinical Treatment (ACT)
Brief Title: A Precision Medicine Approach (SMMART-ACT) for the Treatment of Patients With Advanced Sarcoma, Prostate, Breast, Ovarian or Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Eli Lilly and Company (Industry); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Charles D Lopez, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00026643; NCI-2024-07664 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00026643 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2024-09-26; First posted 2024-10-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Advanced Breast Carcinoma; Advanced Malignant Solid Neoplasm; Advanced Ovarian Carcinoma; Advanced Pancreatic Carcinoma; Advanced Prostate Carcinoma; Advanced Sarcoma; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms | interventions — abemaciclib; Biopsy; Carboplatin; exemestane; Fulvestrant; Gefitinib; Gemcitabine; Letrozole; olaparib; osimertinib; Paclitaxel; Taxes; liposomal doxorubicin; Doxorubicin; Pemetrexed; Tamoxifen; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Arm I (abemaciclib, gemcitabine) (Experimental): Patients receive abemaciclib PO BID on days 1-21 and gemcitabine IV over 30 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.
  Interventions: Drug: Abemaciclib; Procedure: Biopsy; Procedure: Bone Scan; Drug: Gemcitabine; Other: Survey Administration; Procedure: Biospecimen Collection
- Arm II (abemaciclib, pemetrexed) (Experimental): Patients receive abemaciclib PO BID on days 1-21 and pemetrexed IV over 10 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.
  Interventions: Drug: Abemaciclib; Procedure: Biopsy; Procedure: Bone Scan; Drug: Pemetrexed; Other: Survey Administration; Procedure: Biospecimen Collection
- Arm III (abemaciclib) (Experimental): Patients receive abemaciclib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.
  Interventions: Drug: Abemaciclib; Procedure: Biopsy; Procedure: Bone Scan; Other: Survey Administration; Procedure: Biospecimen Collection
- Arm IV (abemaciclib, exemestane) (Experimental): Patients receive abemaciclib PO BID and exemestane PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.
  Interventions: Drug: Abemaciclib; Procedure: Biopsy; Procedure: Bone Scan; Drug: Exemestane; Other: Survey Administration; Procedure: Biospecimen Collection
- Arm V (abemaciclib, letrozole) (Experimental): Patients receive abemaciclib PO BID and letrozole PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.
  Interventions: Drug: Abemaciclib; Procedure: Biopsy; Procedure: Bone Scan; Drug: Letrozole; Other: Survey Administration; Procedure: Biospecimen Collection
- Arm VI (abemaciclib, tamoxifen) (Experimental): Patients receive abemaciclib PO BID and tamoxifen PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.
  Interventions: Drug: Abemaciclib; Procedure: Biopsy; Procedure: Bone Scan; Other: Survey Administration; Drug: Tamoxifen; Procedure: Biospecimen Collection
- Arm VII (gefitinib, pemetrexed, carboplatin) (Experimental): Patients receive gefitinib PO QD on days 1-21, pemetrexed IV on day 1 of each cycle and carboplatin IV on day 1 of cycles 1-6. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.
  Interventions: Procedure: Biopsy; Procedure: Bone Scan; Drug: Carboplatin; Drug: Gefitinib; Drug: Pemetrexed; Other: Survey Administration; Procedure: Biospecimen Collection
- Arm VIII (olaparib, temozolomide) (Experimental): Patients receive olaparib PO BID and temozolomide PO QD on days 1-7 of each cycle. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.
  Interventions: Procedure: Biopsy; Procedure: Bone Scan; Drug: Olaparib; Other: Survey Administration; Drug: Temozolomide; Procedure: Biospecimen Collection
- Arm IX (fulvestrant) (Experimental): Patients receive fulvestrant IM on days 1, 15 and 29 of cycle 1 and day 1 of subsequent cycles. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.
  Interventions: Procedure: Biopsy; Drug: Fulvestrant; Other: Survey Administration; Procedure: Biospecimen Collection
- Arm X (gefitinib) (Experimental): Patients receive gefitinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.
  Interventions: Procedure: Biopsy; Procedure: Bone Scan; Drug: Gefitinib; Other: Survey Administration; Procedure: Biospecimen Collection
- Arm XI (olaparib) (Experimental): Patients receive olaparib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.
  Interventions: Procedure: Biopsy; Procedure: Bone Scan; Drug: Olaparib; Other: Survey Administration; Procedure: Biospecimen Collection
- Arm XII (olaparib, carboplatin, paclitaxel) (Experimental): Patients receive olaparib PO BID on days 1-3, 8-10, 15-17, 21-23 and carboplatin IV and paclitaxel IV on days 1, 8 and 15 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study, as clinically indicated, and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.
  Interventions: Procedure: Biopsy; Procedure: Bone Scan; Drug: Carboplatin; Drug: Olaparib; Drug: Paclitaxel; Other: Survey Administration; Procedure: Biospecimen Collection
- Arm XIII (olaparib, liposomal doxorubicin) (Experimental): Patients receive olaparib PO BID on days 1-28 and liposomal doxorubicin IV on day 1 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography or MUGA scan and blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.
  Interventions: Procedure: Biopsy; Procedure: Bone Scan; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Drug: Olaparib; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Other: Survey Administration; Procedure: Biospecimen Collection
- Arm XIV (osimertinib) (Experimental): Patients receive osimertinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography or MUGA scan and blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.
  Interventions: Procedure: Biopsy; Procedure: Bone Scan; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Drug: Osimertinib; Other: Survey Administration; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY 2835219; LY-2835219; LY2835219; Verzenio
  Arms: Arm I (abemaciclib, gemcitabine); Arm II (abemaciclib, pemetrexed); Arm III (abemaciclib); Arm IV (abemaciclib, exemestane); Arm V (abemaciclib, letrozole); Arm VI (abemaciclib, tamoxifen)
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
  Arms: Arm I (abemaciclib, gemcitabine); Arm II (abemaciclib, pemetrexed); Arm III (abemaciclib); Arm IV (abemaciclib, exemestane); Arm V (abemaciclib, letrozole); Arm VI (abemaciclib, tamoxifen); Arm VII (gefitinib, pemetrexed, carboplatin); Arm VIII (olaparib, temozolomide); Arm X (gefitinib); Arm XI (olaparib); Arm XII (olaparib, carboplatin, paclitaxel); Arm XIII (olaparib, liposomal doxorubicin); Arm XIV (osimertinib)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm VII (gefitinib, pemetrexed, carboplatin); Arm XII (olaparib, carboplatin, paclitaxel)
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
  Arms: Arm XIII (olaparib, liposomal doxorubicin); Arm XIV (osimertinib)
Drug: Exemestane — Given PO
  Other Names: Aromasin; FCE-24304
  Arms: Arm IV (abemaciclib, exemestane)
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ICI-182780; ICI182780; ZD 9238; ZD-9238; ZD9238
  Arms: Arm IX (fulvestrant)
Drug: Gefitinib — Given PO
  Other Names: Iressa; ZD 1839; ZD-1839; ZD1839
  Arms: Arm VII (gefitinib, pemetrexed, carboplatin); Arm X (gefitinib)
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
  Arms: Arm I (abemaciclib, gemcitabine)
Drug: Letrozole — Given PO
  Other Names: CGS 20267; CGS-20267; CGS20267; Femara; Fempro
  Arms: Arm V (abemaciclib, letrozole)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
  Arms: Arm XIII (olaparib, liposomal doxorubicin); Arm XIV (osimertinib)
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
  Arms: Arm VIII (olaparib, temozolomide); Arm XI (olaparib); Arm XII (olaparib, carboplatin, paclitaxel); Arm XIII (olaparib, liposomal doxorubicin)
Drug: Osimertinib — Given PO
  Other Names: AZD 9291; AZD-9291; AZD9291; Mereletinib
  Arms: Arm XIV (osimertinib)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm XII (olaparib, carboplatin, paclitaxel)
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; Pegylated Liposomal Doxorubicin; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
  Arms: Arm XIII (olaparib, liposomal doxorubicin)
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
  Arms: Arm II (abemaciclib, pemetrexed); Arm VII (gefitinib, pemetrexed, carboplatin)
Other: Survey Administration — Ancillary studies
Drug: Tamoxifen — Given PO
  Other Names: TMX
  Arms: Arm VI (abemaciclib, tamoxifen)
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
  Arms: Arm VIII (olaparib, temozolomide)
Procedure: Biospecimen Collection — Biological Sample Collection, Biological Sample Collection, Biospecimen Collected, Biospecimen Collection, Specimen Collection

SUMMARY:
This phase II trial tests the how well a precision medicine approach (serial measurements of molecular and architectural response to therapy [SMMART])-adaptive clinical treatment [ACT]) works in treating patients with sarcoma, prostate, breast, ovarian or pancreatic cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). SMMART testing uses genetic and protein tests to learn how cancer changes and to understand what drugs may work against a person's cancer or why drugs stop working. These test results are reviewed by a group of physicians and scientists during a SMMART tumor board who then recommend precision therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Feasibility of utilizing a SMMART-adaptive clinical treatment (ACT) tumor board to select personalized advanced cancer treatment plans based on a pre-determined set of drug agents with recommended phase 2 doses (RP2Ds).

SECONDARY OBJECTIVES:

I. Safety and tolerability of assigned ACT intervention per cancer type. II. Preliminary indications of efficacy based on disease-specific responses. III. Estimated survival benefit per cancer type.

EXPLORATORY OBJECTIVES:

I. Durability of response compared to the most recent therapy on which progression occurred.

II. Changes in ability to conduct activities of daily living (ADL). III. Changes in quality of life (QoL).

IV. Feasibility of SMMART-centric assessments of ongoing responses to treatment to identify mechanisms of therapy induced change, per investigator discretion. Such mechanisms may include, but will not be limited to, the following:

IVa. Changes in tumor and tumor ecosystem biology; IVb. Response and resistance to therapy.

OUTLINE: Patients are assigned to 1 of 14 arms. Participants may re-enter the study and receive a new arm assignment in the event of progressive disease or unacceptable toxicity.

ARM I: Patients receive abemaciclib orally (PO) twice per day (BID) on days 1-21 and gemcitabine intravenously (IV) over 30 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.

ARM II: Patients receive abemaciclib PO BID on days 1-21 and pemetrexed IV over 10 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.

ARM III: Patients receive abemaciclib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.

ARM IV: Patients receive abemaciclib PO BID and exemestane PO once per day (QD) on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.

ARM V: Patients receive abemaciclib PO BID and letrozole PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.

ARM VI: Patients receive abemaciclib PO BID and tamoxifen PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.

ARM VII: Patients receive gefitinib PO QD on days 1-21, pemetrexed IV on day 1 of each cycle and carboplatin IV on day 1 of cycles 1-6. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment.

ARM VIII: Patients receive olaparib PO BID and temozolomide PO QD on days 1-7 of each cycle. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.

ARM IX: Patients receive fulvestrant intramuscularly (IM) on days 1, 15 and 29 of cycle 1 and day 1 of subsequent cycles. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.

ARM X: Patients receive gefitinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.

ARM XI: Patients receive olaparib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy, CT scan, MRI scan, PET scan and/or bone scan and blood sample collection throughout the study. Additionally, prostate cancer patients undergo bone scan on study.

ARM XII: Patients receive olaparib PO BID on days 1-3, 8-10, 15-17, 21-23 and carboplatin IV and paclitaxel IV on days 1, 8 and 15 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study, as clinically indicated, and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.

ARM XIII: Patients receive olaparib PO BID on days 1-28 and liposomal doxorubicin IV on day 1 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography or multigated acquisition (MUGA) scan and blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.

ARM XIV: Patients receive osimertinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography or MUGA scan and blood sample collection throughout the study. Patients also undergo tumor biopsy on study and optionally at the end of treatment. Additionally, prostate cancer patients undergo bone scan on study.

After completion of study treatment, patients are followed up 30 days, every 3 months for 1 year then every 6 months until year 5.

ELIGIBILITY:
Inclusion Criteria:

* PRE-SCREENING: Written informed consent prior to any Pre-Screening activities, study-specific procedures or interventions
* PRE-SCREENING: At least 18 years of age at time of informed consent. Persons of all gender identities, biological sexes, races, and ethnicities will be included
* PRE-SCREENING: A diagnosis of advanced sarcoma or advanced prostate, breast, ovarian, or pancreatic cancer. Change in an individual's cancer can be tracked objectively according to the Prostate Cancer Working Group 3 (PCWG3) criteria for prostate cancer, and Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 criteria for sarcomas and breast, ovarian, and pancreatic cancers
* PRE-SCREENING: Biospecimen collection, as per institutional standards, must be consented to and collection must be feasible, with the following exceptions for tissue collections:

  * Individuals with a prior tumor tissue sample with successful SMMART-Clinical Analytics Platform (CAP) assays, collected within the last 90 days, may be eligible, so long as ≤ 1 treatment has been received within ≤ 90 days of that biopsy
* PRE-SCREENING: Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* PRE-SCREENING: Physician-assessed life expectancy of ≥ 6 months
* PRE-SCREENING: Additional eligibility criteria specific to their disease must also be met
* PRIMARY TREATMENT: Documented progression after at least 1 line of prior therapy for advanced disease. If recurrence occurred within 6 months of the last dose of an adjuvant/neoadjuvant therapy, that adjuvant/neoadjuvant therapy will count as 1 line of therapy
* PRIMARY TREATMENT: SMMART-ACT tumor board recommendation of at least one SMMART-ACT therapy regimen defined within this protocol, based on the board's review of SMMART-CAP results on a pre-screening biopsy
* PRIMARY TREATMENT: Absolute neutrophil count (ANC) ≥ 1,500/uL (1.5 K/cu mm) (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)
* PRIMARY TREATMENT: Platelets ≥ 100,000/uL (100 K/cu mm) (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)
* PRIMARY TREATMENT: Hemoglobin ≥ 9 g/dL (or ≥ 5.6 mmol/L) (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)
* PRIMARY TREATMENT: Creatinine OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) ≤ 1.5 x institutional upper limit of normal (ULN) (institutional upper limit of normal [IULN]) OR ≥ 50 mL/min/1.73 m^2 (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)

  * Creatinine clearance should be calculated per institutional standard. For participants with a baseline calculated creatinine clearance below normal institutional laboratory values, a measured baseline creatinine clearance should be determined. Individuals with higher values felt to be consistent with inborn errors of metabolism will be considered on a case-by-case basis.
  * Creatinine clearance of > 30 mL/min may be considered given that renal toxicity is not at increased risk and excretion is not major route of clearance for any chosen SMMART-ACT therapeutic
* PRIMARY TREATMENT: Total bilirubin ≤ 1.5 x IULN OR direct bilirubin ≤ IULN for individuals with total bilirubin levels > 1.5 x IULN (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)
* PRIMARY TREATMENT: Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/ Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x IULN (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)
* PRIMARY TREATMENT: International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN, unless individual is receiving anticoagulant therapy, as long as PT or partial thromboplastin time (PTT) is within intended therapeutic range of intended anticoagulant therapy (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)
* PRIMARY TREATMENT: Activated partial thromboplastin time (aPTT) or PTT ≤ 1.5 x ULN, unless participant is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended anticoagulant therapy (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)
* PRIMARY TREATMENT: Body mass index (BMI) > 16.0 and < 35.0 kg/m^2 (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)

  * Participants with a BMI of ≥ 30.0 will use ideal body weight indices in calculating the delivery of agents that are dosed based upon body surface area (i.e., mg agent/meter squared) or weight (i.e., mg agent/kg body weight)
* PRIMARY TREATMENT: Toxicities due to prior therapies should be resolved to baseline or grade 1 (per Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0) before administration of study intervention. The following exceptions are permitted:

  * Alopecia, fatigue, and lymphopenia due to prior therapies.
  * Toxicities attributed to prior anti-cancer therapy that are not expected to resolve and to result in long lasting sequelae (e.g., neuropathy after platinum-based therapy), may be permitted
* PRIMARY TREATMENT: Palliative radiation therapy completed ≥ two weeks prior to start of SMMART-ACT treatment to a measurable disease lesion(s)
* PRIMARY TREATMENT: Study intervention-specific eligibility criteria for the intended, recommended therapy must also be met
* CANCER-SPECIFIC CRITERIA (BREAST CANCER): Lesion(s) remain measurable after systemic therapies, as follows:

  * At least one prior line of pharmacological therapy for hormone receptor (HR) positive, human epidermal growth factor receptor 2 (HER2)-negative disease.
  * At least one prior line of targeted therapy for HER2-positive disease
  * At least one prior line of combination therapy for triple negative disease lacking a BRCA1/2 mutation.
  * At least one prior line of therapy with a PARP inhibitor for triple negative disease with a BRCA1/2 mutation

Exclusion Criteria:

* PRE-SCREENING: Evidence of active malignancy of another cancer with a natural history or treatment history that may affect safety or efficacy assessments of this study or impose unacceptable risk to the participant. Guiding examples for those who can be enrolled include: individuals who have been disease free for ≥ two years; cancers with high cure rates (e.g., prior history of stage 1 rectal cancer and currently otherwise disease free); adequately treated, localized nonmelanomatous skin cancer
* PRE-SCREENING: Absence of biopsiable lesion, AND unavailable/insufficient archival tissue
* PRIMARY TREATMENT: Any brain/central nervous system (CNS) metastasis that progresses within ≤ four weeks of CNS directed treatment as ascertained by clinical examination(s) and MRI or CT during the main eligibility screening period
* PRIMARY TREATMENT: One or more new, active brain/CNS metastasis or the presence of known leptomeningeal disease (LMD) that requires immediate treatment. If treatment within the first cycle of therapy is unlikely to be required, enrollment may be considered, as per the investigator
* PRIMARY TREATMENT: Concurrent forms of anti-cancer therapy that have the potential to interfere with efficacy and safety assessments or that may pose increased risk to the participant while on a SMMART-ACT treatment, and as per the investigator (Select hormone therapies are allowed)
* PRIMARY TREATMENT: More than one intervening line of therapy for treatment of their cancer since the time of the pre-screening biopsy, exclusive of most maintenance hormone therapies

  * Note: Participants who have a pre-screening biopsy while receiving a standard of care (SOC) treatment will not be eligible if they receive any additional lines of treatment prior to the start of SMMART-ACT treatment. This treatment will count as one line of intervening therapy
* PRIMARY TREATMENT: Untreated and/or uncured hepatitis C virus (HCV) infection, as evidenced by detectable hepatitis B core (HBC) ribonucleic acid (RNA) by polymerase chain reaction (PCR). Prior treatment, concurrent treatment, and natural resolution of HCV infection are not exclusionary given (1) no risk for hepatic decompensation and (2) the intended SMMART-ACT treatment is not expected to exacerbate HCV infection
* PRIMARY TREATMENT: Uncontrolled intercurrent illness and infection that may interfere with planned treatment, including, but not limited to, the following:

  * Symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV),
  * Unstable angina pectoris or coronary angioplasty, or stenting within < six months prior to enrollment,
  * Cardiac arrhythmia (ongoing cardiac dysrhythmias of grade ≥ 2 [National Cancer Institute (NCI) CTCAE v 5.0]),
  * Conditions that require intra-cardiac defibrillators,
  * Known cardiac metastases,
  * History of abnormal cardiac valve morphology (≥ grade 2),
  * Chronic graft versus host disease (GVHD) or immunosuppressive therapy for the control of GVHD
* PRIMARY TREATMENT: Severe infection within < four weeks prior to initiation of study therapy, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* PRIMARY TREATMENT: Inability or unwillingness to take oral medication (only for assigned oral study interventions)
* PRIMARY TREATMENT: History of allergy to an assigned study agent or its excipients
* PRIMARY TREATMENT: Current pregnancy, current breastfeeding, or unwillingness to not breastfeed while receiving study drug(s) or for the minimum required time after the last dose of study drug(s) as specified by the SMMART-ACT drug agents
* PRIMARY TREATMENT: Any condition that, in the opinion of the investigator, could jeopardize the participant's safety or adherence to the study protocol
* CANCER-SPECIFIC CRITERIA (PROSTATE CANCER): If the screening bone scan shows a "superscan" participants will be excluded from participation. This is defined as an intense symmetric activity in the bones and diminished renal parenchymal activity, such that the presence of additional metastases in the future could not be evaluated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who receive an adaptive clinical treatment (ACT) therapy based serial measurements of molecular and architectural responses to therapy (SMMART)-ACT tumor board recommendation | From SMMART-ACT tumor board review to the first dose of ACT study drug per unique treatment regimen. This is expected to take up to approximately 30 days.
  A threshold of the posterior probability rate of 75% will be utilized for declaring feasibility to support the analysis of the primary objective in this pilot.

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) suspected or confirmed as attributed to study therapy | From first dose of study drug to 30 days after last dose of study drug(s). This is expected to be approximately 7 months, but could be shorter if participant stops treatment early for any reason.
  The incidence of TEAEs experienced that are suspected or confirmed as attributable to a study drug or procedure will be tabulated
Rate of treatment discontinuation due to toxicities and/or intolerability | From first dose of study drug to last dose of study drug(s). This is expected to be approximately 6 months, but could be shorter if participant stops treatment early for any reason.
  The incidence of discontinuation from study therapy due to intolerability and/or toxicities will be reported.
Overall response rate (ORR) | At 24 weeks from cycle 1 day 1
  ORR is defined as complete response + partial response. Will be assessed per Response Evaluation Criteria in Solid Tumors (RECIST). An exact 95% confidence interval will be provided.
Progression free survival | From first dose of study drug to first date of documented progression or recurrence (RECIST 1.1), end-of-study, or death due to any cause, whichever occurs first, up to 5 years
  Will be estimated using the Kaplan-Meier method.
Disease specific survival (DSS) | From first dose of study drug to death as a result of the disease, up to 5 years
  Will be estimated using the Kaplan-Meier method. Analysis will also fit DSS and subdistribution hazard models for both DSS death and non-DSS death.
Overall survival | From first dose of study drug to date of death from any cause, up to 5 years
  Will be summarized descriptively using the Kaplan-Meier method. The median and 95% confidence interval will be included in the estimations, if possible.

CONTACTS AND LOCATIONS:
Overall Officials: Charles D Lopez, MD, PhD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States